CLINICAL TRIAL: NCT04031508
Title: Effect of a Parenteral Emulsion With LC-PUFA Omega 3 on Clinical Outcomes, Inflammatory and Oxidative Stress Markers in Neonates With Persistent Pulmonary Hypertension Associated With Congenital Diaphragmatic Hernia
Brief Title: Effect of a Parenteral Emulsion With Omega3 on Neonates With PPHN and CDH
Acronym: CDH-PPHN-N3
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: University of Southampton (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Mariela Bernabe García, Full time researcher, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R-2019-785-044
Record Dates: First submitted 2019-07-08; First posted 2019-07-24 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Hypertension of Newborn; Diaphragm Defect
Keywords: PPHN; Diaphragmatic Hernia; omega 3; DHA and EPA
MeSH Terms: conditions — Hernia, Diaphragmatic | interventions — Fish Oils; SMOFlipid

STUDY DESIGN:
Intervention Model Description: Use of a parenteral emulsion that is used as routine nutrition for newborns but not evaluated for persistent pulmonary hypertension.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The attendant gastroenterologist has a randomized allocation and will indicate the type of emulsion during the recruitment. Each emulsion will be designed as a code A or B. The code for each patient is stored into an opaque envelop, which is opened once the parents have given their written informed consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 (Experimental): The experimental group will receive a parenteral emulsion containing soy oil, MCT, olive oil and n-3 LCPUFA in fish oil
  Interventions: Combination Product: lipid injectable emulsion with Fish oil
- Control group (Sham Comparator): The Control group will receive a parenteral emulsion containing soy oil and MCT
  Interventions: Combination Product: lipid injectable emulsion with Fish oil

INTERVENTIONS:
Combination Product: lipid injectable emulsion with Fish oil — TPN will start at 1.5-2.0 g/kg/d of the lipid emulsion, increasing 1.0 g/kg/d until a maximum of 3.0 g/kg/d for at least 7 days.
  Other Names: SMOFLIPID

SUMMARY:
The purpose of this study is to evaluate the effect of a parenteral emulsion containing n-3 long-chain polyunsaturated fatty acids (LC-PUFA) in fish oil on clinical outcomes, markers of inflammation and oxidative stress, and pain in neonates with persistent pulmonary hypertension of the newborn (PPHN) compared with those who receive an emulsion containing soy oil and medium-chain triglycerides (MCT) without n-3 LC-PUFA.

DETAILED DESCRIPTION:
Background. Persistent pulmonary hypertension of the newborn (PPHN), is a syndrome characterized by difficulty to provide normal pulmonary vasodilatation at birth or after birth, which may be related to right ventricular dysfunction, congenital diaphragmatic hernia, sepsis, and meconium aspiration. This condition is understudied. PPHN causes pulmonary vascular resistance (PVR) that decreases left pulmonary artery flow (LPA), meaning that blood cannot be oxygenated in the lungs, leading to low oxygen delivery to all organs. Expensive medication along with ventilator support may help, but the latter and PPHN increase the production of the inflammatory mediators such as pro-inflammatory cytokines and markers of oxidative stress, which cause cell toxicity. To treat the hernia, infants undergo corrective surgery, which further increases the production of inflammatory markers and worsens oxidative stress. As a result, the pain of the surgery also worsens the hypoxemia and respiratory insufficiency in the newborn. PPHN is associated with chronic lung disease (CLD). To date, there is no effective treatment for neonates with PPHN, and around one-third of patients may not respond to current management, leading to the death of up to 33% of infants in developed countries. In Mexico, the mortality rate from PPHN may reach 80%, which is an unacceptable outcome at a high cost. Therefore, the prevention or reduction of the severity of PPHN is actively sought.

Previous reports have shown that the n-3 long-chain polyunsaturated fatty acids (LC-PUFA), such as docosahexaenoic acid (DHA) improves the nutritional status and clinical outcomes in septic newborn reduce systemic inflammation and organ dysfunction in newborns who underwent cardiovascular surgery with a shorter stay in the neonatal intensive care unit. In addition, those babies received lower amounts of analgesics. Other authors have shown that n-3 LC-PUFA reduces oxidative stress. In experimental models of PPHN, the EPA and DHA from Omegaven (fish oil) increased pulmonary artery flow and decrease pulmonary vascular resistance. In the current project, it is hypothesized that n-3 LC-PUFA improves clinical outcomes such as decreasing pulmonary vascular pressure and markers of inflammation and oxidative stress in neonates with PPHN. This hypothesis has not been evaluated.

Objective. The purpose of this study is to evaluate the effect of a parenteral emulsion containing n-3 LC-PUFA in fish oil on clinical outcomes, markers of inflammation and oxidative stress, and pain in neonates with PPHN compared with those who receive an emulsion containing soy and medium-chain triglycerides (MCT) without n-3 LC-PUFA.

Methodology. A double-blind clinical trial will be carried out on Mexican newborns diagnosed with PPHN. The control group will receive intravenous nutrition support including a lipid emulsion based on soy oil plus MCT (control group) and the intervention group will receive a lipid emulsion based on soy oil, MCT, olive oil, and fish oil (n-3 LC-PUFA group); both groups will receive a dose of lipid (3 g/kg/d maximum), through total parenteral nutrition (TPN) for at least 7 days.

The effect of n-3 LC-PUFA will be evaluated on:

1. Clinical outcomes, nutritional status, the manifestation of pain
2. Markers of inflammation
3. Oxidative stress markers

To compare the groups, the Exact Fisher´s, Student's t, or U-Mann-Whitney tests will be applied as appropriate. To adjust the effect of n-3 LC-PUFA for confounders such as fatty acid background and medication, Repeated Measures ANOVA and binary logistic regression will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Plan to administrate TPN for at least 7 days
* Clinical, gasometric, and echocardiographic diagnosis of congenital diaphragmatic hernia.
* Gestational age >=34 weeks.
* Written informed consent signed by both parents after an explanation of the objectives, procedures and possible risks and benefits of the research, along with the signature of two witnesses

Exclusion Criteria:

* Diagnosis of complex congenital cardiopathy
* Cyanotic congenital cardiology defect
* Insufficiency of the tricuspid valve
* Immunosuppressive disease. HIV has been associated with PPHN and human herpesvirus with vascular remodeling, perivascular macrophages, and lung fibrosis
* Clinical entities that preclude the total parenteral nutrition for one day or longer.
* Presence of profuse and persistent haemorrhage at any level

Elimination criteria

* Parents who withdraw their consent.
* Starting a drug at doses for nonclotting treatment such as heparin, enoxaparin.
* Development of profuse and persistent haemorrhage at any level after receiving vitamin K treatment.

Ages: 1 Hour to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change on systolic pressure of pulmonary artery | Before surgery (baseline), 24 hour, 48 hour, 72 hour, day 7, day 14 and day 21 post-surgery.
  Measured by echocardiography in millimeters of mercury (mm/Hg)
Preductal partial pressure of carbon (PaCO2) | Before surgery (baseline), 24 hour, 48 hour, 72 hour and day 7 post-surgery.
  Good response if the carbon in blood is <60-70 mmHg measured by gasometry in arterial blood
Change in Preductal and postductal oxygen saturation (SatO2) | Before surgery (baseline), 24 hour, 48 hour, 72 hour, day 7, day 14 and day 21 post-surgery.
  It is a measure of oxygenation in hemoglobin. It is preductal if the measurement id on hand, and postductal if it is on foot, determined by an pulse oximeter in percentage
Inspired fraction of oxygen (FiO2) | Before surgery (baseline), 24 hour, 48 hour, 72 hour, day 7, day 14 and day 21 post-surgery.
  Oxygen concentration supplied by ventilation support in percentage
Growth velocity and Nutritional status | Before surgery (baseline), day 7, day 14 and day 21 post-surgery.
  Measurement of body weight in grams, length, and head circumference in centimeters (if clinical condition allows it) to obtain grams/kg/d, cm/week, Z score, and eutrophic or undernutrition outcome using the Fenton's standard reference of growth and/or World Health Organization as appropriate for preterm or term infants, respectively.
Pain manifestation | Before surgery (baseline), 24 hour, 48 hour, 72 hour, day 7, day 14 and day 21 post-surgery.
  Pain will be measured with the COMFORT scale computed by eight sections with scores from 1 to 5 each.

SECONDARY OUTCOMES:
Concentration of plasma cytokines as inflammatory markers | Before surgery (baseline), 24 hour, 48 hour, 72 hour, and day 7 post-surgery.
  Determination of pro and anti-inflammatory cytokines interleukin (IL)-1beta, tumoral necrosis factor-alpha, IL-6, IL-8, IL-10, IL-12 (p70) (pg/milliliter) in plasma by luminex-based immunoassay.
Concentration of inflammatory derived-lipid mediators | Before surgery (baseline), 24 hour, 48 hour, 72 hour, and day 7 post-surgery.
  Determination lipid mediators such as eicosanoids and resolvin(s) in ng/ml by liquid chromatography coupled to mass spectrometry.
Concentration of total free thiols | At study entry, before surgery (2 baselines), and once a day until day 7 after surgery, then at 14 and 21 days-post-surgery.
  This will be measured in urine by ELISA in pg/milliliter
Concentration of nitrotyrosine | At study entry, before surgery (2 baselines), and once a day until day 7 after surgery, then at 14 and 21 days-post-surgery.
  This will be measured in urine by ELISA in micromol per liter (uM)
Concentration of the nuclear factor erythroid 2-related factor 2 (Nrf2) | At study entry, before surgery (2 baselines), and once a day until day 7 after surgery, then at 14 and 21 days-post-surgery.
  This will be measured in urine by ELISA in pg/milliliter
Concentration of Ratio of F2-isoprostanes (F2-isop) and F2-isofurans (F2-isof) | At study entry, before surgery (2 baselines), and once a day until day 7 after surgery, then at 14 and 21 days-post-surgery.
  This ratio will be measured in urine in nmol/liter by Liquid chromatography coupled to mass spectrometry.
Chronic Lung Disease | At hospital discharge or 56 day-old, at 6 months and one year of age
  It will be evaluated with the need of supplementary Oxygen and/or medication to improve lung function

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Bernabe-Garcia, Ph.D., Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unit of Medical Research in Nutrition, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: experimental model report in DOI: 10.1097/CCM.0b013e31821204fb — https://pubmed.ncbi.nlm.nih.gov/21378553/